CLINICAL TRIAL: NCT03219567
Title: Whole Eye Optical Coherence Tomography (OCT) to Improve Refractive Surgery and Eye Care
Status: Terminated | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00056946
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2021-11

CONDITIONS: Image, Body
MeSH Terms: interventions — Tomography, Optical Coherence; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Normals (Experimental): Normal subjects will be imaged with the OCT system to ensure the imaging range of the system.
  Interventions: Device: Optical Coherence Tomography (OCT)
- Patients with a history of cataract surgery or high myopia (Experimental): Subjects will be imaged with both the OCT system and MRI. Reconstructions of the eye from each modality will then be compared.
  Interventions: Device: Optical Coherence Tomography (OCT); Device: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Device: Optical Coherence Tomography (OCT) — Optical coherence tomography (OCT) is a non-contact, micrometer scale imaging technique, it provides clinicians and researchers with high resolution in vivo images sufficient to visualize layered microanatomy in 3D.
  The study team will develop the hardware systems and software algorithms necessary to enable simultaneous OCT imaging of all the refractive surfaces of the eye.
Device: Magnetic resonance imaging (MRI) — Magnetic resonance imaging (MRI) is a medical imaging technique that uses a magnetic field and computer-generated radio waves to create detailed images of the organs and tissues in the body.
  Arms: Patients with a history of cataract surgery or high myopia

SUMMARY:
The overall objective is to develop the hardware systems and software algorithms necessary to make accurate measurements of the whole eye with optical coherence tomography (OCT).

The research procedure that each subject will undergo is imaging with the OCT system. Three populations will be included: 1. Normals to ensure the imaging range of the system, 2. Patients with previous LASIK who will be undergoing cataract surgery, and 3. Patients with a history of cataract surgery or high myopia. The third group will also undergo MRI imaging for comparison.

There are no known risks to the subject from imaging with optical coherence tomography beyond what is normal for standard ocular photographic procedures. Light exposure is below ANSI limits. In groups 2 and 3, clinical parameters drawn from the OCT images will be compared to standard of care imaging.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older.
* Pseudophakic group: has had prior uncomplicated cataract surgery with a monofocal or toric intraocular lens, able to undergo head MRI
* High myopia group: refraction equal to or stronger than -6 D spherical equivalent, able to undergo head MRI

Exclusion Criteria:

* under 21 years of age, unable or unwilling to give consent.
* Pseudophakic group: complications with cataract surgery or insertion of a multifocal intraocular lens, failure to pass MRI pre-screening (e.g. prior metallic implants, claustrophobic), unable to fixate.
* High myopia group: failure to pass MRI pre-screening, unable to fixate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-10-09 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Normals: Normal subjects will be imaged with the OCT system to ensure the imaging range of the system.
  Optical Coherence Tomography (OCT): Optical coherence tomography (OCT) is a non-contact, micrometer scale imaging technique, it provides clinicians and researchers with high resolution in vivo images sufficient to visualize layered microanatomy in 3D.
  The study team will develop the hardware systems and software algorithms necessary to enable simultaneous OCT imaging of all the refractive surfaces of the eye.
- Patients With a History of Cataract Surgery or High Myopia: Subjects will be imaged with both the OCT system and MRI. Reconstructions of the eye from each modality will then be compared.
  Optical Coherence Tomography (OCT): Optical coherence tomography (OCT) is a non-contact, micrometer scale imaging technique, it provides clinicians and researchers with high resolution in vivo images sufficient to visualize layered microanatomy in 3D.
  The study team will develop the hardware systems and software algorithms necessary to enable simultaneous OCT imaging of all the refractive surfaces of the eye.
  Magnetic resonance imaging (MRI): Magnetic resonance imaging (MRI) is a medical imaging technique that uses a magnetic field and computer-generated radio waves to create detailed images of the organs and tissues in the body.
Period: Overall Study
Arm/Group | Normals | Patients With a History of Cataract Surgery or High Myopia
Started | 18 | 64
Completed | 18 | 63
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normals | Patients With a History of Cataract Surgery or High Myopia | Total
Number analyzed (Participants) | 18 | 64 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (12.1) | 73.3 (12.7) | 72.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 21 | 33
  Male | 6 | 43 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 62 | 78
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 15 | 15
  White | 16 | 42 | 58
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 64 | 82

OUTCOME MEASURES:

1. Primary Outcome: Difference in Radius of Curvature (Rc) of the Posterior Eye From OCT Compared to MRI
Description: The radius of curvature of the posterior eye will be measured via surface fitting of the posterior eye data from OCT and MRI. Data reported reflects the Rc of the posterior eye measured by OCT minus the value obtained by MRI measurement.
Time Frame: 36 months
Population: Participants who were imaged with both the OCT system and MRI ("Patients with a history of cataract surgery or high myopia" group only). Data not collected on 40 participants.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Groups:
- Patients With Previous LASIK Who Will be Undergoing Cataract Surgery: Patients with previous LASIK who will be undergoing cataract surgery subjects will be imaged with the OCT system.
  Optical Coherence Tomography (OCT): Optical coherence tomography (OCT) is a non-contact, micrometer scale imaging technique, it provides clinicians and researchers with high resolution in vivo images sufficient to visualize layered microanatomy in 3D.
  The study team will develop the hardware systems and software algorithms necessary to enable simultaneous OCT imaging of all the refractive surfaces of the eye.
Arm/Group | Normals | Patients With Previous LASIK Who Will be Undergoing Cataract Surgery | Patients With a History of Cataract Surgery or High Myopia
Number analyzed (Participants) | 0 | 0 | 42
Number analyzed (eyes) | 0 | 0 | 80
mm |  |  | -0.11 (0.35)
Statistical Analysis 1: Comparison: Patients With a History of Cataract Surgery or High Myopia; OCT compared to MRI; Test type: Other; p = 0.35, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Normals | Patients With a History of Cataract Surgery or High Myopia
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/64
Other Adverse Events (participants affected / at risk) | 0/18 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT03219567/Prot_SAP_000.pdf